CLINICAL TRIAL: NCT04594850
Title: An Single-blind, Multi-center, Randomization, Phase Ⅱ Study to Evaluate Efficacy and Safety of Cellgram-ED (Autologous Bone Marrow-derived Mesenchymal Stem Cells) in Erectile Dysfunction Patients With Following Radical Prostatectomy
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of of Autologous Mesenchymal Stem Cells (MSC) Injected Intracavernously
Acronym: Cellgram-ED
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmicell Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMC-P-10
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo-Control group (No Intervention): Single intracavernous injection of Placebo Oral PDE5-inhibitor can take daily and on demand.
- Injection group: Cellgram-ED (Experimental): Single intracavernous injection of Mesenchymal stem cell. Oral PDE5-inhibitor can take daily and on demand.
  Interventions: Biological: Cellgram-ED

INTERVENTIONS:
Biological: Cellgram-ED — Patients will receive single injection of Cellgram-ED(mesenchymal stem cell) intracavernously.
  Other Names: Autologous bone marrow derived mesenchymal stem cell
  Arms: Injection group: Cellgram-ED

SUMMARY:
This phase II clinical trial is designed to evaluate the efficacy and safety of autologous Mesenchymal Stem Cells (MSC) injected intracavernously.

DETAILED DESCRIPTION:
To evaluate the efficacy and efficacy for 12 months after a single dose of Cellgram-ED in patients with erectile dysfunction after radical prostatectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 19 to 80 years old at screening
2. Patients who maintained normal foot function before prostatectomy and are interested in restoring sexual function after surgery
3. PSA level <10 ng/mL before prostatectomy
4. Pathological Gleason sum ≤ 7(3+4 or 4+3) factor during prostatectomy
5. Local lesions that did not metastasize during prostatectomy (pT2, N0, M0 stage) factors
6. Patients more than 1 year after prostatectomy and PSA ≤ 0.04 ng/mL when screened without additional treatment other than surgery
7. Who cannot satisfy sexual activity(more than 4 times) with proper sexual stimulation in spite of taking maximum dose of oral PDE5I(phos-phodiesterasetype-5 inhibitors) within last 8weeks.
8. Total score of 10 or more and 17 or less in the EF (Erectile function) field* of the International Erectile Function Questionnaire

   * 1, 2, 3, 4, 5, 15 questions for EF erectile function in the international erectile function questionnaire
9. Prevalence for erectile dysfunction at screening with more than 6 months
10. Who are willing to engage in sexual activity more than 4 times a month and have a constant partner for at least 3 months
11. Who do not have difficulty reading and understanding the contents of the questionnaire and who fill out a complete questionnaire
12. A person who voluntarily agrees to participate in this clinical trial and has signed the consent form by the subject and the subject partner

Exclusion Criteria:

1. Severe cardiovascular disease (angina pectoris, myocardial infarction, unstable arrhythmia, heart failure, etc.) at the screening visit
2. Who cannot collect bone marrow due to bone marrow disease, etc.
3. Those with the following medical history/companion diseases A. Gentamicin hypersensitivity reaction B. Solid cancer or malignant blood disease within 5 years prior to screening C. Clinically significant cognitive impairment, dementia or psychiatric disorder D. Alcohol or substance abuse E. Priapism F. Severe respiratory diseases (COPD, asthma, pneumonia, pulmonary embolism, pneumothorax, etc.) G. Stroke H. Systemic autoimmune disease
4. Those with the following test results at the screening visit A. Liver disease or abnormal liver function (AST or ALT ≥ 3 times the normal upper limit of the organ) B. Severe renal impairment (serum creatinine≥ 2 mg/dL) C. Positive factors for pathogenic microbial tests (Hbs Ag, HCV Ab, HIV Ab, Syphilis) D. Uncontrolled high blood pressure (systolic blood pressure >170 mmHg or diastolic blood pressure >100 mmHg) or hypotension (systolic blood pressure <90 mmHg, diastolic blood pressure <50 mmHg) E. Who are outside the normal range of tumor marker tests (PSA, CEA, AFP) F. Hemorrhagic tendency (PT and aPTT> ULN x 1.5) G. Untreated hypogonadism or serum testosterone hormone less than 200 ng/dL
5. Those who possess the following therapeutic powers at screening A. Who are being treated for severe systemic or local infection B. Long-term use of anticoagulant (warfarin) (administered for more than 3 months as anticoagulant therapy) C. Vacuum compressor or intracavernous injection therapy within 7 days before screening (prostaglandin E1, papaverine, phentolamine, etc.) D. Immunosuppressants, alpha blockers or male hormones (androgens, anti-androgens) within 28 days prior to screening
6. Penile anatomical malformations (ex: Peyronie's disease) or penile implants or penile vascular procedures
7. Who are receiving drugs* that are expected to affect the results of this clinical trial when judged by the investigator
8. If the partner is a woman of childbearing potential, those who are not willing to use an appropriate contraceptive method** during the clinical trial period

   **Contraceptive administration and implantation or intrauterine device, infertility procedures (vapectomy, tubal ligation, etc.), blocking method (condom, contraceptive diaphragm, vaginal sponge or cervical cap)
9. Who participated in other interventional clinical trials within 4 weeks prior to the screening visit and received clinical investigational drugs/investigational medical devices or received procedures
10. Who have or will be administered other cell therapy products
11. A person who is judged to be inappropriate to participate in this test when judged by the examiner

Random Inclusion Criteria:

1. Total score of 10 or more and 17 or less in the EF (Erectile function) field* of the International Erectile Function Questionnaire (IIEF)

   * 1, 2, 3, 4, 5, 15 questions for EF erectile function in the international erectile function questionnaire
2. Who attempts sexual activity more than 4 times during the run-in period and has a failure rate (Sexual Encounter Profile) of 50% or more

Ages: 19 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2026-01-07 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
The amount of change in EF score in the International Erectile Function Questionnaire (IIEF) at administration of the clinical trial drug compared to the baseline value | 6 month
  Descriptive statistics for the amount of change at administration of the investigational drug compared to the baseline value for each administration group are presented and analyzed by an analysis of covariance (ANCOVA)
  Erectile Function (Q1,2,3,4,5,15) : Min 6 ~ Max 30 Orgasmic Function (Q9,10) : Min 2 ~ Max 10 Sexual Desire (Q11,12) : : Min 2 ~ Max 10 Intercourse Satisfaction (Q6,7,8): : Min 3 ~ Max 15 Overall Satisfaction (Q13,14) : Min 2 ~ Max 10

SECONDARY OUTCOMES:
The amount of change in EF score in the International Erectile Function Questionnaire (IIEF) at administration of the clinical trial drug compared to the baseline value | month 1, 3, 6, 9 and 12
  Descriptive statistics for the amount of change at administration of the investigational drug compared to the baseline value for each administration group are presented and analyzed by an analysis of covariance (ANCOVA)
  Erectile Function (Q1,2,3,4,5,15) : Min 6 ~ Max 30
Changes in SEP Q 2 and Q 3 evaluation after administration of investigational drug compared to baseline | month 1, 3, 6, 9 and 12
  Descriptive statistics for the success rate change at each time point and baseline value for each administration group are presented and analyzed by covariance analysis (ANCOVA)
  SEP 2 Were you able to insert your penis into your partner's vagina? Yes or No SEP 3 Did your erection last long enough to have successful intercourse? Yes or No
Global Assessment Question (GAQ) evaluation after administration of investigational drugs | month 1, 3, 6, 9 and 12
  The frequency and percentage of each time point by administration group are presented and analyzed by Pearson's chi-square test or Fisher's exact test
  Did Cellgram-ED improve your Erectile Function? Yes or No If so, did Cellgram-ED improve the ability to have sex? Yes or No
Changes in Penile Doppler Sonography(PDS) level after administration of clinical trial drug compared to baseline | month 6, 12
  For the continuous variable, descriptive statistics for each time point in each administration group and the change at each time point compared to the baseline value are presented, and analyzed by covariance analysis (ANCOVA)
  PDS results are obtained 5 min, 10 min, 15 min, 20 min, 25 min and 30 min after intracavernosal injection.
  The peak systolic velocity (PSV) is assessed as follows: >25 cm/s is considered to be normal, 20-25 cm/s is considered to be mild ED, 12-20 cm/s is considered to be moderate ED, <12 cm/s is considered to be severe arteriogenic impotence.
  The end diastolic velocity (EDV) is assessed as follows: 5 cm/s is considered to be a normal value, >5 cm/s is considered to indicate a veno-occlusive disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Chungsu Kim, Ph.D, Principal Investigator — AIDS Malignancy Consortium
Locations (4):
- South Korea (4):
  - Asan medical center, Seoul
  - Ewha womans university medical center, Seoul
  - Samsung medical center, Seoul
  - Seoul ST. Mary's hospital, Seoul